CLINICAL TRIAL: NCT00824616
Title: A Phase IIa, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial of MK-0941 in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Insulin
Brief Title: A Study to Test MK-0941 in Adults With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on Insulin (MK-0941-018)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0941-018; 2009_516 (Other: Merck Registration ID); MK-0941-018 (Other: Merck Protocol ID)
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-((6-(ethylsulfonyl)-3-pyridinyl)oxy)-5-(2-hydroxy-1-methylethoxy)-N-(1-methyl-1H-pyrazol-3-yl)benzamide; Insulin; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Participants receiving placebo tablets three times daily plus insulin injection once daily
  Interventions: Drug: Placebo; Drug: Insulin
- MK-0941 (Experimental): Participants receiving MK-0941 tablets three times daily plus insulin injection once daily
  Interventions: Drug: MK-0941; Drug: Insulin

INTERVENTIONS:
Drug: MK-0941 — MK-0941 tablets 5 mg or 10 mg, taken 3 times daily, with increasing doses to maximally effective dose.
  Arms: MK-0941
Drug: Placebo — Placebo tablets, taken 3 times daily.
  Arms: Placebo
Drug: Insulin — Insulin glargine (rDNA origin) injection solution for subcutaneous (SC) injection, taken once daily.
  Other Names: LANTUS®

SUMMARY:
The purpose of this study is to test the effect MK-0941 as add-on therapy for adults taking insulin for Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participant has Type 2 Diabetes Mellitus

Exclusion Criteria:

* Participant has a history of Type 1 Diabetes Mellitus or ketoacidosis
* Participant is on a weight loss program and is not in the maintenance phase or is taking a weight loss medication
* Participant has had surgery within 30 days of starting the study or has planned major surgery

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants receiving Placebo tablets 3 times daily plus insulin injection once daily
- MK-0941: Participants receiving MK-0941 tablets 3 times daily plus insulin injection once daily
Period: Overall Study
Arm/Group | Placebo | MK-0941
Started | 34 | 34
Completed | 28 | 27
Not Completed | 6 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Creatinine/Creatinine Clearance | 0 | 2
Not completed — Hyperglycemia | 1 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MK-0941 | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (8.8) | 54.1 (10.2) | 54.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) Level
Description: HbA1c level is a blood test measurement of the amount (percent) of hemoglobin that is glycated (or has glucose on it). HbA1c level is related to the average blood glucose concentration over the previous 2-3 months, with a higher HbA1c level indicating a higher amount of average plasma glucose. A negative number for change from baseline in HbA1c level means a reduction in HbA1c level and indicates better control of average plasma glucose levels.
Time Frame: Baseline (Day 1) and End of Treatment (Week 20)
Population: Full Analysis Set Population, which consisted of all randomized participants who took at least one dose of study drug (MK-0941 or Placebo) and had a baseline or post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: % HbA1c
Arm/Group | Placebo | MK-0941
Number analyzed (Participants) | 34 | 34
% HbA1c | -0.15 [-0.65 to 0.34] | -0.26 [-0.76 to 0.23]
Statistical Analysis 1: Comparison: Placebo vs MK-0941; Test type: Superiority or Other; p = 0.745, Longitudinal Data Analysis (LDA) model; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.81 to 0.58]

2. Primary Outcome: Number of Participants Who Experienced One or More Episodes of Hypoglycemia (Symptomatic or Asymptomatic)
Description: Hypoglycemic episodes - with or without symptoms - are defined as a fingerstick glucose measurement of ≤70 mg/dL (3.9 mmol/L). Excludes data after initiation of glycemic rescue therapy.
Time Frame: From first dose of study drug (Week 0) to last dose of study drug (Week 20)
Population: All Participants as Treated Population, which consisted of all randomized participants who took at least one dose of study drug (MK-0941 or Placebo).
Measure: Number; unit: participants
Arm/Group | Placebo | MK-0941
Number analyzed (Participants) | 34 | 34
participants | 6 | 8
Statistical Analysis 1: Comparison: Placebo vs MK-0941; Between-treatment difference (MK-0941 group minus Placebo group) in the percentage of participants who experienced one or more episodes of hypoglycemia; Test type: Superiority or Other; p = 0.537, Miettinen & Nurminen method; Proportions = 5.9, 95% CI 2-sided [-13.7 to 25.4]

ADVERSE EVENTS:
Time Frame: From Screening Visit 2 (Week -10) through to 2 weeks after last dose of randomized study drug (up to 32 weeks)
Description: Reporting of serious AEs includes data after initiation of glycemic rescue therapy. Reporting of non-serious AEs excludes data after initiation of glycemic rescue therapy.
Arm/Group | Placebo | MK-0941
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/34
Other Adverse Events (participants affected / at risk) | 13/34 | 11/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | MK-0941 (N=34)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | MK-0941 (N=34)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (9) | 8 (50)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After multicenter publication or 24 months after study completion, whichever comes first, an investigator may publish the results for their study site only. Sponsor can review publications 60 days prior to submission.